CLINICAL TRIAL: NCT04491305
Title: Implementation of Endometriosis Health Profile-5 (EHP-5) in Croatian Gynecological Practice for Preoperative Assessment in Women With Endometriosis
Brief Title: EHP-5 in Preoperative Assessment in Women With Endometriosis
Acronym: EHP-5CRO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Zagreb (Other)
Responsible Party: Principal Investigator, Mislav Mikuš, MD, University of Zagreb
Other Study IDs: PetrovaZg
Record Dates: First submitted 2020-07-25; First posted 2020-07-29 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Endometriosis; Endometriosis Ovary; Endometriosis-related Pain; Quality of Life; Endometrioma; Endometriosis, Rectum
Keywords: endometriosis; quality of life
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with pathohistological confirmation: Women aged between 18 and 50 with surgically proven endometriosis.
  Interventions: Procedure: Surgically treated women with endometriosis and confirmed diagnosis

INTERVENTIONS:
Procedure: Surgically treated women with endometriosis and confirmed diagnosis — Women with indication for surgery or diagnostic laparoscopy will be enrolled in study.

SUMMARY:
There is no validated tool in quality-of-life assessment of women with endometriosis in Croatia. First aim is to validate Endometriosis Health Profile-5 (EHP-5) before implementing this questionnaire in clinical practice. After validation, we will prospectively follow women with endometriosis through whole process - pre- and postoperatively.

DETAILED DESCRIPTION:
There is no validated tool in quality-of-life assessment of women with endometriosis in Croatia. First aim is to validate Endometriosis Health Profile-5 (EHP-5) before implementing this questionnaire in clinical practice. After validation, we will prospectively follow women with endometriosis through whole process - pre- and postoperatively, including comparison with rASRM and Enzian score which are already established in our Clinic.

We will try to identify correlation between EHP-5 score and surgical findings and to provide better insight in quality of life consideration of women with endometriosis particularly in Croatia. Since we are tertiary referral centre with almost 250 operative procedures which include ovarian, pelvic and/or extra pelvic endometriosis, we believe that this study will bring new tool not only for preoperative assessment but postoperative surveillance.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 50 years; symptoms of endometriosis (pelvic pain, dyspareunia, dysmenorrhea) for at least 6 months or previously verified primary sterility; pathohistological confirmation of diagnosis after surgical treatment or indicated diagnostic laparoscopy; fluent and literate in Croatian language; ability to independently understand the questions in the questionnaires

Exclusion Criteria:

* pregnant women; cognitive impairment or intellectual disability; neurological disorders (e.g. epilepsy, Parkinson disease, multiple sclerosis, cerebrovascular insult); lack of independent mobility and polytraumatic patients; diagnosed vulvodynia and active vulvovaginitis; ongoing urinary tract infection; any form of prior conservative and/or surgical treatment for endometriosis; lack of informed consent

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: We will include at least 100 women with surgically proven endometriosis in order to establish EHP-5 in our clinical practice.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
EHP-5 score can predict extent of surgical procedure | Intraoperative time
  Bigger overall EHP-5 score will be successful predictor of required surgical intervention

SECONDARY OUTCOMES:
EHP-5 score in postoperative surveillance | Postoperative routine surveillance at two different time points - 6 weeks and 6 months after operation
  We assume that EHP-5 score can be used as a postoperative surveillance indicator

CONTACTS AND LOCATIONS:
Overall Officials: Mislav Mikuš, MD, Principal Investigator — University Hospital Center Zagreb, Croatia
Locations (1):
- Clinical Hospital Centre Zagreb, Croatia, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No